CLINICAL TRIAL: NCT06732960
Title: A Randomized, Double-Blind, Placebo-controlled Study of Efsubaglutide Alfa on Weight Management in Subjects With Overweight or Obesity to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics, and Efficacy.
Brief Title: A Study of the Efficacy and Safety of Efsubaglutide Alfa in Overweight or Obesity Patients
Acronym: LIGHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Yinnuo Pharmaceutical Technology Co., Ltd. (Other)
Collaborators: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Beijing Friendship Hospital (Other); Jinan Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: YN011-W201; YN011-W201 (Other: Guangzhou Innogen Pharmaceutical Group Co., Ltd.)
Record Dates: First submitted 2024-12-05; First posted 2024-12-13 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-12

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Efsubaglutide Alfa 5mg (Experimental): 10 eligible subjects will be randomized in a 8:2 manner to receive either Efsubaglutide Alfa or Placebo, Dose escalation of Efsubaglutide Alfa or Placebo should take place during the first 4 weeks after randomization as describe in detail description. All subjects should aim at reaching the recommended target dose of Efsubaglutide Alfa 5 mg once-weekly maintenances 4 weeks or the corresponding volume of Placebo.
  Interventions: Biological: Efsubaglutide Alfa; Other: Placebo
- Efsubaglutide Alfa 7.5mg (Experimental): 10 eligible subjects will be randomized in a 8:2 manner to receive either Efsubaglutide Alfa or Placebo, Dose escalation of Efsubaglutide Alfa or Placebo should take place during the first 4 weeks after randomization as describe in detail description. All subjects should aim at reaching the recommended target dose of Efsubaglutide Alfa 7.5 mg once-weekly maintenances 4 weeks or the corresponding volume of Placebo.
  Interventions: Biological: Efsubaglutide Alfa; Other: Placebo
- Efsubaglutide Alfa 10mg (Experimental): 10 eligible subjects will be randomized in a 8:2 manner to receive either Efsubaglutide Alfa or Placebo, Dose escalation of Efsubaglutide Alfa or Placebo should take place during the first 6 weeks after randomization as describe in detail description. All subjects should aim at reaching the recommended target dose of Efsubaglutide Alfa 10 mg once-weekly maintenances 4 weeks or the corresponding volume of Placebo.
  Interventions: Biological: Efsubaglutide Alfa; Other: Placebo
- Efsubaglutide Alfa 15mg (Experimental): 10 eligible subjects will be randomized in a 8:2 manner to receive either Efsubaglutide Alfa or Placebo, Dose escalation of Efsubaglutide Alfa or Placebo should take place during the first 8 weeks after randomization as describe in detail description. All subjects should aim at reaching the recommended target dose of Efsubaglutide Alfa 10 mg once-weekly maintenances 4 weeks or the corresponding volume of Placebo.
  Interventions: Biological: Efsubaglutide Alfa; Other: Placebo
- Efsubaglutide Alfa 20mg (Experimental): 10 eligible subjects will be randomized in a 8:2 manner to receive either Efsubaglutide Alfa orPlacebo, Dose escalation of Efsubaglutide Alfa or Placebo should take place during the first 12 weeks after randomization as describe in detail description. All subjects should aim at reaching the recommended target dose of Efsubaglutide Alfa 10 mg once-weekly maintenances 4 weeks or the corresponding volume of Placebo.
  Interventions: Biological: Efsubaglutide Alfa; Other: Placebo

INTERVENTIONS:
Biological: Efsubaglutide Alfa — Efsubaglutide Alfa subcutaneous injection under 1mg, 3mg, 5mg, 7.5mg, 10mg, 15mg or 20mg dose weekly.
  Other Names: Supaglutide
Other: Placebo — Placebo subcutaneous injection weekly

SUMMARY:
This is a study to evaluate the safety, efficacy, pharmacokinetics and pharmacodynamics of Efsubaglutide Alfa at difference dose range once-weekly in patients with Overweight or Obesity.

DETAILED DESCRIPTION:
This study will look at the adverse events and the change in participants' body weight from the start of the study to the end. Weight loss in participants taking Efsubaglutide Alfa will be compared to weight loss in participants taking placebo.

ELIGIBILITY:
Inclusion Criteria:

* Fully understood the study, signed the informed consent.
* Male or female patients aged from 18 to 75 years at the time of signing informed consent.
* Body mass index (BMI) greater than or equal to 28 kg/sqm or greater than or equal to 24 kg/sqm with the presence of at least one of the following weight-related comorbidities: prediabetic state, hypertension, dyslipidemia, non-alcoholic steatohepatitis (NASH), obstructive sleep apnea or cardiovascular disease.
* A self-reported change in body weight less than 5% within 90 days before screening irrespective.

Exclusion Criteria:

* Glycated hemoglobin (HbA1c) greater than or equal to 6.5%, or previously diagnosed with type 1 diabetes or type 2 diabetes.
* Have history of clinically significant abnormal gastric emptying, severe chronic gastrointestinal diseases, long-term use of medications that directly affect gastrointestinal peristalsis, or gastrointestinal surgery within 6 months prior to screening, and deemed unsuitable for participation by the investigator.
* Have history of hyperthyroidism or hypothyroidism, or a thyroid-stimulating hormone (TSH) level below the lower limit or above 1.5 times the upper limit of the normal range.
* Calcitonin greater than or equal to 50 ng/L, or have history of medullary thyroid carcinoma, multiple endocrine neoplasia (MEN) type 2A or 2B syndrome, or a related family history.
* Any other condition that, in the judgment of the researchers, may affect the patient's ability to provide informed consent or comply with the trial protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-04-21 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Weight | Baseline, 4 weeks after the target dose
  Relative Change in Body Weight (%), Proportion of subjects with a weight loss of ≥5% from baseline
Adverse Event | Adverse events occurring within 4 weeks of the last dose from baseline
  Numbers of Adverse Event

SECONDARY OUTCOMES:
Weight | Baseline, 4 weeks after the target dose
  Proportion of subjects with a weight loss of ≥10% or ≥15% from baseline, Change from baseline in weight
BMI | Baseline, 4 weeks after the target dose
  Change from baseline in BMI
Waist circumference | Baseline, 4 weeks after the target dose
  Change from baseline in Waist circumference
Hip circumference | Baseline, 4 weeks after the target dose
  Change from baseline in Hip circumference
Waist Hip Rate (WHR) | Baseline, 4 weeks after the target dose
  Change from baseline in Waist Hip Rate (WHR)
Diastolic pressure | Baseline, 4 weeks after the target dose
  Change from baseline in Diastolic pressure
Systolic pressure | Baseline, 4 weeks after the target dose
  Change from baseline in Systolic pressure
Triglyceride | Baseline, 4 weeks after the target dose
  Change from baseline in Triglyceride
Total Cholesterol | Baseline, 4 weeks after the target dose
  Change from baseline in Total Cholesterol
High Density Lipoprotein Cholesterol （HDL-C） | Baseline, 4 weeks after the target dose
  Change from baseline in High Density Lipoprotein Cholesterol （HDL-C）
Low-Density Lipoprotein Cholesterol （LDL-C） | Baseline, 4 weeks after the target dose
  Change from baseline in Low-Density Lipoprotein Cholesterol （LDL-C）
HbA1c | Baseline, 4 weeks after the target dose
  Change from baseline in HbA1c
Fasting Blood Insulin | Baseline, 4 weeks after the target dose
  Change from baseline in Fasting Blood Insulin
HOMA-IR | Baseline, 4 weeks after the target dose
  Change from baseline in HOMA-IR
Body Fat | Baseline, 4 weeks after the target dose
  Change in body fat from baseline measured with a body fat scale.

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Jia, M.D,Ph. D, Principal Investigator — Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Locations (3):
- China (3):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, China
  - Jinan Central Hospital Affiliated to Shandong First Medical University, Jinan, China
  - Shanghai Sixth People's Hospital Affiliated to Shanghai JiaoTong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No